CLINICAL TRIAL: NCT06093789
Title: The Relationship Between Personality Traits and Perioperative Anesthetic Drug Consumption
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, SEZGİN BİLGİN, MD, Ondokuz Mayıs University
Other Study IDs: PT-PADC
Record Dates: First submitted 2023-07-10; First posted 2023-10-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Infertility
Keywords: Personality traits; Anesthetic Drug Consumption; Anxiety; Acute pain
MeSH Terms: conditions — Infertility; Anxiety Disorders; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group PT-PADC: patients who will receive sedoanalgesia for the oocyte retrieval procedure.
  Interventions: Other: PBQ-S1

INTERVENTIONS:
Other: PBQ-S1 — All patients will fill out Personality Belief Scale-Short Form (PBQ-S1) and Beck Anxiety Scale one day before the procedure and they will be registered.

SUMMARY:
In this study, we aimed to examine the association between personality traits and amount of anesthetic drug consumption,of the patients who will receive sedoanalgesia for the oocyte retrieval procedure. As well as determining the anxiety scores in the preoperative period, the time to reach the desired sedation level, hemodynamic parameters in the perioperative period, peripheral oxygen saturation, EtCO2 value, postoperative pain, postanesthetic recovery, analgesic drug need, unconscious movement, and patient satisfaction.

DETAILED DESCRIPTION:
Different personality traits, anxiety disorders, depression, and somatoform disorders are frequently encountered in women with infertility problems. Although there are many studies evaluating the relationship of anxiety with variables such as hemodynamic parameters, need for anesthetic medication, recovery times, postoperative pain and analgesic requirements, the relationship between personality traits and these variables has not been investigated.

In our study, considering that the anesthesia needs of these patients with a stressful negative factor such as infertility may be at different levels, preoperative evaluation of the patients with a personality questionnaire will provide better perioperative management, a better quality recovery and possibly a higher quality oocyte aspiration. In this study, it was aimed to investigate the amount of anesthetic agent consumption, recovery times, postoperative pain scores, analgesic requirements, involuntary movement, time to reach sufficient sedation depth, and patient satisfaction of patients thought to have sedation.

All patients will fill out Personality Belief Scale-Short Form (PBQ-S1) and Beck Anxiety Scale one day before the procedure and they will be registered.

ELIGIBILITY:
Inclusion Criteria:

* 18- 50 year-old elective patients who signed the informed consent form from ASA I-II patients scheduled for oocyte retrieval.
* Patients with sufficient education and mental capacity to complete in assessment scales and questionnaires.
* Patients without neurological disorders, psychological illnesses, or drug or alcohol abuse
* Patients without stimulant drug and alcohol consumption
* Absence of significant cardiovascular, respiratory, kidney or liver disease.

Exclusion Criteria:

* Psychiatric or neurological disorder
* Psychiatric drug use or alcohol consumption
* Pregnancy
* Presence of severe cardiac, hepatic or cerebrovascular disease
* History of allergy to local anesthetics or systemic opioids
* History of chronic pain
* Patients who are unable to evaluate scales and questionnaires

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Female patients between 18-50 ages who will undergo oocyte pick up procedure with sedation
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Propofol consumption | from the beginning to the end of the transvaginal oocyte retrieval procedure)
  mg, from the beginning to the end of the transvaginal oocyte retrieval procedure

SECONDARY OUTCOMES:
Time until the Ramsey Sedation Score of 4 is reached | -The period of time starting with the propofol injection until the Ramsey Sedation Score of 4
  The period elapsed after the patient is transported to the operating table and the sedation protocol begins.
Amount of propofol (mg) used until the required sedation depth is reached | The period of time starting with the propofol injection until the Ramsey Sedation Score of 4
  The amount of iv propofol administered until the Ramsey Sedation Score of 4 is obtained
Systolic, diastolic and, mean Blood pressure (mm/Hg) | every 5 minutes during the procedure
  It will be monitored and documented every 5 minutes during the procedure.
Heart rate (beats/min) | every 5 minutes during the procedure.
  It will be monitored and documented every 5 minutes during the procedure.
Peripheral oxygen saturation (%) | every 5 minutes during the procedure
  (%): It will be monitored and documented every 5 minutes during the procedure.
Number of Involuntary movement during the procedure | during the procedure.
  The presence of involuntary movement will be documented during the procedure.
Postoperative pain (visual analog scale) | After the procedure,every 30 minutes up to 1 hour
  Pain status will be evaluated based on visual analog scale (VAS) at rest and after movement.every 30-minute intervals for one hour in the recovery room. Each VAS is scores 0-10 (0=no pain, 10=unbearable pain)
Analgesic consumption | postoperatively up to 2 hours
  The analgesic agents administered to the patients throughout the postoperative period will be documented.
Postoperative recovery time | postoperatively up to 2 hours
  The time until the Modified Aldrete Score reaches 9 points will be determined.
The incidences of post-operative nausea and vomiting (PONV) | the time from the end of the procedure until discharge
  the presence of nausea and vomiting will be recorded for 24 hours after procedure
Undesirable events and interventions | time between start of procedure and discharge
  Bradycardia, hypotension, airway obstruction, hypoxia will be documented throughout the perioperative phase with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Lee SS, Kim HH, Park HJ. Are Histrionic Personality Traits Associated with Irritability during Conscious Sedation Endoscopy? Gastroenterol Res Pract. 2015;2015:702492. doi: 10.1155/2015/702492. Epub 2015 Apr 12. PMID 25954307
- [Background] Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 1999 Dec;89(6):1346-51. doi: 10.1097/00000539-199912000-00003. PMID 10589606
- [Background] CLARIDGE GS, HERRINGTON RN. Sedation threshold, personality, and the theory of neurosis. J Ment Sci. 1960 Oct;106:1568-83. doi: 10.1192/bjp.106.445.1568. No abstract available. PMID 13693809